CLINICAL TRIAL: NCT00321503
Title: Diagnosis and Response to Treatment of Laryngopharyngeal Reflux Using an Oropharyngeal Aerosolized pH Probe
Brief Title: Study of an Oropharyngeal Aerosolized pH Probe for Diagnosing Laryngopharyngeal Reflux (LPR)
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: AstraZeneca (Industry); Respiratory Technology Corporation (Industry)
Responsible Party: Principal Investigator, Adam Klein, Principal Investigator, Emory University
Other Study IDs: 1345-2005; DX-1 for LPR (Other: other)
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Laryngopharyngeal Reflux
Keywords: acid reflux; LPR; gastroesophageal reflux; GERD; pH probe; proton pump inhibitor; PPI
MeSH Terms: conditions — Laryngopharyngeal Reflux; Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study is a test of how well a new FDA-approved device is for diagnosing a condition known as laryngopharyngeal reflux (LPR). The device, which measures pH of the air in the upper throat, will be compared to several other methods for diagnosing laryngopharyngeal reflux.

DETAILED DESCRIPTION:
It is estimated that up to 50% of patients with voice disorders and 4-10% of patients seen in otolaryngology practice experience laryngopharyngeal reflux (LPR). LPR has been implicated in the pathogenesis of numerous laryngeal disorders, including subglottic stenosis, laryngeal carcinoma, laryngeal contact ulcers, laryngospasm, and vocal cord nodules. In the pediatric population, it has been associated with asthma, sinusitis, and otitis media. Common symptoms include chronic and intermittent hoarseness, vocal fatigue, globus pharyngeus, cough, postnasal drip, chronic throat clearing, and dysphagia.

Like gastroesophageal reflux disease (GERD), the etiology of LPR is linked to esophageal sphincter dysfunction. In GERD, the lower esophageal sphincter (LES) is involved, whereas in LPR, the pathology results from upper esophageal sphincter (UES) dysfunction. However, diagnosis of LPR is more challenging than that of GERD. The classic reflux-like symptoms of heartburn and regurgitation are often absent in LPR.

The most widely used diagnostic modality for LPR is symptomatic response to treatment, including twice daily proton pump inhibitor (PPI) or H2 blocker therapy for several months. However, the use of a therapeutic modality to make a diagnosis clearly carries disadvantages, including potentially unnecessary exposure to a drug's side effect profile and lengthy time to diagnosis. Another diagnostic instrument is the reflux symptom index (RSI), a validated nine-item questionnaire assessing LPR symptoms. However, LPR symptoms are fairly nonspecific, also appearing in autoimmune and behavior disorders. Lastly, a 24-hour triple-pH probe may be the best objective test diagnosing LPR. However, this method is poorly tolerated by patients and difficulty with ease of administration limits its routine use. To date, we have remained in search of a minimally invasive and specific test for LPR.

In this study, we will investigate the use of a newly developed oropharyngeal pH probe for detecting aerosolized acid as an accurate and minimally invasive diagnostic instrument for LPR. This device has previously been shown to correlate to lower esophageal, upper esophageal, and lower pharyngeal pH as measured by a 24-hour triple channel bifurcated pH probe [ACG Poster session by Dr. G Wiener]. The number of oropharyngeal aerosolized acid reflux events and acid exposure times will be compared to RSI before and after twice daily proton pump inhibitor therapy. In addition, the correlation between acid reflux events and acid exposure times as measured by the Dx probe will be more rigorously compared to that measured by a triple pH probe.

ELIGIBILITY:
INCLUSION CRITERIA:

Group 1 (negative control):

* RSI ≤ 13
* No history of voice or swallowing disorders
* No active voice or swallowing disorders
* No history of heartburn, regular indigestion, and no prior or current diagnosis of GERD

Groups 2 and 3 (experimental group):

* Clinical symptoms consistent with LPR as measured by an RSI > 13.
* No other voice or swallowing pathology on clinical exam

EXCLUSION CRITERIA:

* Regular treatment with an H2 blocker or proton pump inhibitor (PPI)
* History of laryngeal/pharyngeal surgery
* Any planned treatment of the larynx/pharynx other than treatment for LPR
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pos controls: Subjects visiting the Emory Clinic/Emory Voice center with LPR symptoms.
  Neg controls: Random subjects in Atlanta without LPR symptoms. See other descriptions for more details.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Klein, MD, Principal Investigator — Dept of Otolaryngology; Michael M Johns, MD, Study Chair — Dept of Otolaryngology / Director of Emory Voice Center; Leena Khaitan, MD, MPH, Principal Investigator — Dept of Surgery; Justin S Golub, BA, Study Director — Emory University
Locations (1):
- Emory Voice Center, Atlanta, Georgia, United States

REFERENCES:
- [Background] Belafsky PC, Postma GN, Koufman JA. Validity and reliability of the reflux symptom index (RSI). J Voice. 2002 Jun;16(2):274-7. doi: 10.1016/s0892-1997(02)00097-8. PMID 12150380
- [Background] Merati AL, Lim HJ, Ulualp SO, Toohill RJ. Meta-analysis of upper probe measurements in normal subjects and patients with laryngopharyngeal reflux. Ann Otol Rhinol Laryngol. 2005 Mar;114(3):177-82. doi: 10.1177/000348940511400302. PMID 15825565